CLINICAL TRIAL: NCT04641650
Title: FreeStyle Libre Pro Flash Continuous Glucose Monitoring (CGM) System in Subjects With Diabetes on HemoDIALsis (FSL-DIAL Pilot Study)
Brief Title: Pilot Study : FreeStyle Libre Pro Flash Continuous Glucose Monitoring System in Subjects With Diabetes on HemoDIALsis
Acronym: FSL DIAL
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Saint Joseph Saint Luc de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: FSL DIAL
Record Dates: First submitted 2020-11-18; First posted 2020-11-24 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Kidney Failure; Diabetes
Keywords: glycemia; diabetes; kidney failure; dialysis; glucose sensor
MeSH Terms: conditions — Renal Insufficiency; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Continuous monitoring of glucose with a FreeStyle Libre pro sensor in diabetic and dialysis patients

ELIGIBILITY:
Inclusion Criteria:

* Diabetes without any change in treatment in the last 3 months
* Hemodialysis for > 3 months
* Recent laboratory HbA1c (< 15 days)

Exclusion Criteria:

* Patient does not show non-opposition
* Skin allergy to the sensor
* Sepsis / Acute anaemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with diabetes on hemodialysis
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2022-11-09 (Actual); Study Completion 2022-11-09 (Actual)

PRIMARY OUTCOMES:
Difference between estimated Hba1c (or Glucose Management Index (GMI)) with FreeStyle Libre Pro sensor and laboratory Hba1c | At sensor removal (day 14)
  Comparison between estimated HbA1c with 14 days of CGM data and laboratory HbA1c (routine blood test in hemodialysis) in each subject

SECONDARY OUTCOMES:
Time in glucose range | At sensor removal (day 14)
  Percent (%) time in glucose range of ≥70 to ≤180 mg/dL (≥3.9 to ≤10 mmol/L), obtained using professional continuous glucose monitoring (CGM)
Time with Glucose < 70mg/dL | At sensor removal (day 14)
  % time with glucose <70 mg/dL
Time with Glucose > 180 mg/dL | At sensor removal (day 14)
  % time with glucose >180 mg/dL
Glucose total coefficient of variation (CV) | At sensor removal (day 14)
  Glucose total CV (%)

CONTACTS AND LOCATIONS:
Overall Officials: Lucien Marchand, MD, Principal Investigator — Study Principal Investigator
Locations (1):
- Centre Hospitalier Saint Joseph Saint Luc, Lyon, France

IPD SHARING:
Plan to Share IPD: No